CLINICAL TRIAL: NCT02115880
Title: PRimary Prevention Of Depression in Offspring of Depressed Parents
Acronym: PRODO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Bavarian State Ministry of Environment, Public Health and Consumer Protection (Other Government)
Responsible Party: Principal Investigator, Professor Gerd Schulte-Körne, Prof. Dr., Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LP00216_PRODO; LP00216 (Other Grant/Funding Number: Bavarian State Ministry of Environment, Public Health and Consumer Protection)
Record Dates: First submitted 2014-04-07; First posted 2014-04-16 (Estimated); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Depression
Keywords: Depression; Prevention; Adolescent; Child; Randomised Controlled Trial; Risk; Cognitive behavioural therapy; Group-based therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prevention programme (Experimental)
  Interventions: Behavioral: Prevention programme
- Control (treatment as usual) (No Intervention)

INTERVENTIONS:
Behavioral: Prevention programme — Based on a group- and family-based cognitive behavioural manual developed by Bruce Compas and colleagues in the USA, and adapted for a German sample. The programme is for parents and children and consists of 8 weekly sessions and 4 monthly booster sessions.
  Arms: Prevention programme

SUMMARY:
The purpose of this randomised controlled trial is to see whether a group-based psychological intervention for families can reduce the inflated risk of depression in children and adolescents who have at least one parent who suffers from depression (or who has suffered from depressed in the child's lifetime).

ELIGIBILITY:
Inclusion Criteria:

* At least one parent who meets diagnostic criteria for a current (or past, during the child's lifetime) diagnosis of depression
* The participating child is aged 8-17
* The participating child has an IQ of at least 85
* Both child and parent(s) have adequate German-language skills
* Both child and parents consent to intervention sessions being video-recorded

Exclusion Criteria:

* The participating parent(s) has current symptoms of bipolar disorder, psychotic symptoms, personality disorder, substance addiction, or is suicidal
* The participating child meets criteria for a current, or previous, episode of any psychiatric disorder
* The participating child is undergoing or has undergone treatment for depression
* The participating child or parent have serious symptoms of a disorder (or are in crisis) that may hamper their ability to take part in the study

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2014-05; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Presence or absence of a depressive episode (child) | T4 (9 months after completion of the programme)
  The German version of the Diagnostic Interview for Psychiatric Disorders in Children and Adolescents (Kinder DIPS) will be used to assess whether the child meets the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for a depressive episode.

SECONDARY OUTCOMES:
Symptoms of depression (child) | Within 2 weeks of the last session of the intervention (T2) as well as 3 months after the intervention (T3) and 9 months after the intervention (T4)
  Self-reported symptoms of depression will be collected using the German questionnaires "Depression Inventory for Children and Adolescents" (DIKJ) and Beck Depression Inventory (BDI-II; depending on the child's age).
Psychopathological symptoms (child) | Within 2 weeks of the last session of the intervention (T2) as well as 3 months after the intervention (T3) and 9 months after the intervention (T4)
  More general internal and external psychopathological symptoms will be measured using German versions of the questionnaires "Youth Self-Report" (YSR; child self-report) and "Child Behaviour Checklist" (CBCL; parent-report).

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Schulte-Körne, MD, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Department of Child and Adolescent Psychiatry, Psychosomatics, and Psychotherapy, Munich, Bavaria, Germany

REFERENCES:
- [Background] Compas BE, Forehand R, Thigpen JC, Keller G, Hardcastle EJ, Cole DA, Potts J, Watson KH, Rakow A, Colletti C, Reeslund K, Fear J, Garai E, McKee L, Merchant MJ, Roberts L. Family group cognitive-behavioral preventive intervention for families of depressed parents: 18- and 24-month outcomes. J Consult Clin Psychol. 2011 Aug;79(4):488-99. doi: 10.1037/a0024254. PMID 21707137
- [Background] Compas BE, Forehand R, Keller G, Champion JE, Rakow A, Reeslund KL, McKee L, Fear JM, Colletti CJ, Hardcastle E, Merchant MJ, Roberts L, Potts J, Garai E, Coffelt N, Roland E, Sterba SK, Cole DA. Randomized controlled trial of a family cognitive-behavioral preventive intervention for children of depressed parents. J Consult Clin Psychol. 2009 Dec;77(6):1007-20. doi: 10.1037/a0016930. PMID 19968378
- [Derived] Lochner J, Platt B, Starman-Wohrle K, Takano K, Engelmann L, Voggt A, Loy F, Bley M, Winogradow D, Hammerle S, Neumeier E, Wermuth I, Schmitt K, Oort F, Schulte-Korne G. A randomized controlled trial of a preventive intervention for the children of parents with depression: mid-term effects, mediators and moderators. BMC Psychiatry. 2023 Jun 21;23(1):455. doi: 10.1186/s12888-023-04926-2. PMID 37344778
- [Derived] Lochner J, Starman-Wohrle K, Takano K, Engelmann L, Voggt A, Loy F, Bley M, Winogradow D, Hammerle S, Neumeier E, Wermuth I, Schmitt K, Oort F, Schulte-Korne G, Platt B. A randomised controlled trial of a family-group cognitive-behavioural (FGCB) preventive intervention for the children of parents with depression: short-term effects on symptoms and possible mechanisms. Child Adolesc Psychiatry Ment Health. 2021 Oct 1;15(1):54. doi: 10.1186/s13034-021-00394-2. PMID 34598737
- [Derived] Claus N, Marzano L, Loechner J, Starman K, Voggt A, Loy F, Wermuth I, Haemmerle S, Engelmann L, Bley M, Schulte-Koerne G, Platt B. Qualitative evaluation of a preventive intervention for the offspring of parents with a history of depression. BMC Psychiatry. 2019 Sep 18;19(1):290. doi: 10.1186/s12888-019-2273-6. PMID 31533676
- [Derived] Platt B, Pietsch K, Krick K, Oort F, Schulte-Korne G. Study protocol for a randomised controlled trial of a cognitive-behavioural prevention programme for the children of parents with depression: the PRODO trial. BMC Psychiatry. 2014 Sep 18;14:263. doi: 10.1186/s12888-014-0263-2. PMID 25269863
- See also: Related Info — http://www.kjp.med.uni-muenchen.de/forschung/prodo.php